CLINICAL TRIAL: NCT03038529
Title: Variable Approaches of Intradiscal O3-O2 Injection for Management of Low Back Pain: Could it Make a Difference? a Prospective Double Blind Randomized Clinical Trial.
Brief Title: Variable Approaches of Intradiscal O3-O2 Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Lecturer of Anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00009903
Record Dates: First submitted 2017-01-28; First posted 2017-01-31 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Low Back Pain
Keywords: low back pain , Ozone
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: Classic approach (Other): Intradiscal O3 injection through classic postrolateral extraarticular percutaneous approach.
  The participants will receive 10 ml of ozone oxygen mixture 30 ug O3/ml O2. The ozone-oxygen mixture was produced in real-time by a medical ozone generator (Ozonline E 80, Medica srl, Bologna Italy).
  Interventions: Procedure: Classic postrolateral extraarticular percutaneous approach for O3 injection
- B: Transforaminal approach (Yess approach ) (Active Comparator): Participants will receive 10 ml of ozone oxygen mixture 30 ug O3/ml O2 through postrolateral transforaminal approach (Yess approach).
  The ozone-oxygen mixture was produced in real-time by a medical ozone generator (Ozonline E 80, Medica srl, Bologna Italy).
  Interventions: Procedure: Postrolateral transforaminal approach (Yess approach ) for O3 injection

INTERVENTIONS:
Procedure: Classic postrolateral extraarticular percutaneous approach for O3 injection — Receive 10 ml of ozone oxygen mixture 30 ug O3/ml O2 through the classic postrolateral extraarticular percutaneous approach
  Arms: A: Classic approach
Procedure: Postrolateral transforaminal approach (Yess approach ) for O3 injection — Group B receive 10 ml of ozone oxygen mixture 30 ug O3/ml O2 through postrolateral transforaminal approach (Yess approach ).
  Arms: B: Transforaminal approach (Yess approach )

SUMMARY:
Cost Intradiscal injection of ozone-oxygen mixture (O3-O2) which offers a rapid onset amelioration of symptoms, with a sustained duration pain relief in low back pain.

Does change of injection approach make a difference?

DETAILED DESCRIPTION:
Low back pain (LBP) mostly is induced by disc herniation (DH), or degeneration and has a burden upon social and economic aspects of life. Medical and or surgical interventions have been used to resolve this problem, but one of the newly introduced is the minimally invasive low cost Intradiscal injection of ozone-oxygen mixture (O3-O2) which offers a rapid onset amelioration of symptoms, with a sustained duration pain relief.

A lot of injection approaches are available, but which offers the best results, is the question.

ELIGIBILITY:
Inclusion Criteria:

* radicular leg pain
* low back pain
* non-responsive to conservative treatment

Exclusion Criteria:

* patient refusal
* infection at injection site
* coagulopathy
* uncontrolled or degenerative spine disease
* pregnancy
* multilevel disk involvement

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Quality of pain alleviation (visual analog scale) | one year
  assessing visual analog scale (VAS)

SECONDARY OUTCOMES:
Analgesia reduction (percent) | one year
  the percent of analgesia reduction

CONTACTS AND LOCATIONS:
Overall Officials: Abdelraheem Alawaamy, MD, Study Director — Assiut University
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided